CLINICAL TRIAL: NCT06017648
Title: Prospective, Multicenter, Randomized, Blinded, Parallel-Controlled Trial on the Efficacy and Safety of the Focused Ultrasound Device (FUBA5200) for Noninvasive Fat Reduction
Brief Title: A Multicenter Controlled Study to Evaluate Efficacy and Safety of Focused Ultrasound Device (FUBA5200) for Noninvasive Fat Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Carnation Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HJ002-07-001
Record Dates: First submitted 2023-08-21; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Body Sculpting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group 1 - Non Invasive Ultrasound (FUBA5200) (Experimental): Treatment with the Focused Ultrasound Fat Reduction device (FUBA5200) 4 times in total, once every two weeks
  Interventions: Device: Non Invasive Ultrasound (FUBA5200)
- Active comparator: Group 2 - Non Invasive Ultrasound (Contour I V3) (Active Comparator): Treatment with the focused ultrasound fat reduction device (Contour I V3) 4 times in total, once every two weeks
  Interventions: Device: Non Invasive Ultrasound (Contour I V3)

INTERVENTIONS:
Device: Non Invasive Ultrasound (FUBA5200) — the Focused Ultrasound Fat Reduction device (FUBA5200) is manufactured by Shanghai Carnation Medical Technology Co., Ltd
  Arms: Experimental: Group 1 - Non Invasive Ultrasound (FUBA5200)
Device: Non Invasive Ultrasound (Contour I V3) — the Focused Ultrasound Fat Reduction device (Contour I V3) is manufactured by Syneron Medical Ltd.
  Arms: Active comparator: Group 2 - Non Invasive Ultrasound (Contour I V3)

SUMMARY:
This clinical trial is a prospective, multicenter, randomized blinded, parallel controlled study. The purpose of this study is to evaluate the efficacy and safety of the Focused UltrasoundDevice (FUBA5200) for Fat Reduction.

DETAILED DESCRIPTION:
This clinical trial is a prospective, multicenter, randomized blinded, parallel controlled study. The purpose of this study is to evaluate the efficacy and safety of the Focused UltrasoundDevice (FUBA5200) for Fat Reduction.The primary objective of this study is to evaluate the effectiveness of the FUBA5200 System on abdominal circumference reduction at last visit relative to active comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~55 years;
2. Abdominal fat thickness of at least 2.0 cm;
3. Body mass index (BMI) <28.0 kg/m2;
4. Simple localized obesity with abdominal subcutaneous fat accumulation;
5. Those who voluntarily participate in this clinical trial and sign informed consent, agreeing to maintain the same dietary and exercise habits during the study period as before treatment, and to maintain changes in body weight of no more than ±6%;
6. For women of childbearing potential with negative serum pregnancy tests at Screening/baseline;
7. Those who have not participated in any clinical trials within three months prior to enrollment.

Exclusion Criteria:

1. Pregnant women, breastfeeding women or women at childbearing age who are expected to become pregnant or who are prone to contraceptive failure;
2. Subjects with pacemakers, implantable cardiac defibrillators or other electromagnetic implantable medical systems;
3. History of underlying medical conditions such as hypertension (blood pressure ≥ 140/90 mmHg), hyperlipidemia, diabetes, hyperthyroidism or hypothyroidism;
4. Patients who are positive for 4 preoperative infection tests (including anti-human immunodeficiency virus antibodies, syphilis spirochete-specific antibodies, hepatitis C virus antibodies, and hepatitis B surface antigen, in which any one of these is positive);
5. Patients with autoimmune or connective tissue diseases or malignant tumors;
6. Those with cardiac, hepatic or renal insufficiency (Alanine aminotransferase or Aspartate Transaminase > 1.5 times the upper limit of normal; Blood urea nitrogen > 1.5 times the upper limit of normal or Cr > the upper limit of normal; ischemic heart disease; cardiac valvular disease; congestive heart failure);
7. Abnormal coagulation, abnormal blood counts, and dyslipidemia (total cholesterol, triglycerides, or LDL exceeding 20% of the upper limit of the normal range);
8. History of exposure to high fat-soluble compounds (e.g., pesticides, herbicides, or drugs known to be stored in fat, except oral contraceptives), use of retinoids within the last 1 month;
9. History of lacerations or dermatologic conditions, active dermatologic conditions, known tendency to form keloids or poor wound healing in the area of treatment; current infectious lesions in the area of treatment and its immediate vicinity;
10. Abdominal hernia, diastasis recti or known abdominal aortic aneurysm (abdominal treatment);
11. History of fat reduction procedures at the treatment site (e.g., undergoing liposuction, surgery, use of lipolytic agents, etc.) or history of other surgeries or presence of implants at the required treatment site and its adjacent areas;
12. Non-invasive or minimally invasive fat reduction, skin tightening, or lipolysis treatments such as ultrasound, radiofrequency, etc., on the abdomen within the past 6 months;
13. Received weight loss treatment methods (including medication, physical therapy and controlled diet and exercise therapy) within the past 1 month;
14. Those who are allergic to medical device treatments and excipients and acoustic gel for this treatments;
15. Concomitant use with anti-aggregating drugs (non-steroidal anti-inflammatory drugs NSAIDS, etc.). o) Concomitant use with anticoagulant drugs (Warfarin, etc.);
16. Subjects with unrealistic expectations of therapeutic efficacy;
17. Patients with legally defined disabilities (blindness, deafness, dumbness, mental retardation, physical disability);
18. Persons with mental disorders;
19. Patients who are unable or unwilling to comply with the requirements of the study;
20. Subject is in other conditions deemed unsuitable for the trial by the investigator judgment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Reduction in circumference measurement of the abdomen from baseline | Week 10
  The primary objective of this study is to evaluate the effectiveness of the FUBA5200 System on abdominal circumference reduction at last visit relative to active comparator (last visit (visit 7)：28 days after the 4th treatment).

SECONDARY OUTCOMES:
Reduction in circumference measurement of the abdomen every visit | Day 0、1 and week 2、4、6
  The second objective of this study is to evaluate the effectiveness of the FUBA5200 System on abdominal circumference reduction of abdomen every visit (visit 2, 3, 4, 5 and 6).
Assess abdominal subcutaneous fat thickness reduction from baseline to the last visit | Week 10
  evaluate the effectiveness of the FUBA5200 System on abdominal subcutaneous fat thickness reduction of abdomen at visit 7.
Assess subject satisfaction measured with a self-assessment questionnaire (Likert scale) | Week 10
  Subject satisfaction with FUBA5200 as determined by the results of a subjects satisfaction questionnaire at the visit 7. Subject satisfaction was designed as a 5-level standard (0-5)，the higher the level, the higher the satisfaction.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing
  - Huashan Hospital Fudan University, Shanghai